CLINICAL TRIAL: NCT03147066
Title: Efficacy of Dezocine for the Prevention of Catheter-related Bladder Discomfort
Brief Title: Dezocine for Prevention of Catheter-related Bladder Discomfort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jian-jun Yang (Other)
Responsible Party: Sponsor-Investigator, Jian-jun Yang, Director, Department of Anesthesiology, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20170110
Record Dates: First submitted 2017-05-02; First posted 2017-05-10 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-08

CONDITIONS: Catheter Related Bladder Discomfort
Keywords: Dezocine; CRBD; General anesthesia; Urinary catheter
MeSH Terms: interventions — dezocine; flurbiprofen axetil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dezocine (Experimental): 0.1 mg/kg of intravenous dezocine 30 min before the end of surgery
  Interventions: Drug: Dezocine
- Flurbiprofen axetil (Active Comparator): 1 mg/kg of intravenous flurbiprofen axetil 30 min before the end of surgery
  Interventions: Drug: Flurbiprofen Axetil

INTERVENTIONS:
Drug: Dezocine — Dezocine (0.1 mg/kg）will be infused during surgery
  Other Names: Dalgan
  Arms: Dezocine
Drug: Flurbiprofen Axetil — Flurbiprofen Axetil (1 mg/kg）will be infused during surgery
  Arms: Flurbiprofen axetil

SUMMARY:
This study evaluates the efficacy of dezocine in preventing the catheter-related bladder discomfort (CRBD) in a postanesthesia care unit (PACU).

DETAILED DESCRIPTION:
Thirty min before the end of the surgery, patients were randomly assigned to one of the two group to receive intravenous dezocine 0.1 mg/kg (Group D, n=48) or flurbiprofen axetil 1 mg/kg (Group F, n=48) . The CRBD was assessed at 0, 1, 2, and 6 h after patient's arrival in the post-anaesthesia care unit. Severity of CRBD was graded as none, mild, moderate and severe.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>/=18)
2. Male or female
3. Patients scheduled for abdominal surgery
4. Undergoing catheterization
5. Subject is American Society of Anesthesiologists (ASA) physical status 1 or 2

Exclusion Criteria:

1. Patient with bladder outflow obstruction
2. Patient with overactive bladder (frequency greater than three times per night or more than eight times per 24 h)
3. Patient with multisystemic diseases (central nervous system, cardiovascular system hepatic, psychiatric, and end-stage renal diseases)
4. Patient with chemical substance abuse
5. Patient with chronic pain
6. Patient with morbid obesity
7. Patient needs for urgent intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Catheter related bladder discomfort symptoms | at 1 hour after extubatio
  CRBD will be evaluated with a 4 point scale (1; no discomfort, 2; mild, revealed on questioning only, 3; moderate, stated by the patient without questioning, 4; severe, urinary urgency executed by behavioral responses, such as attempts to remove urinary catheter, restless extremity movements, verbal responses)

SECONDARY OUTCOMES:
Catheter related bladder discomfort symptoms | at 0, 1, 2, and 6 hours after extubation
  CRBD will be evaluated with a 4 point scale (1; no discomfort, 2; mild, revealed on questioning only, 3; moderate, stated by the patient without questioning, 4; severe, urinary urgency executed by behavioral responses, such as attempts to remove urinary catheter, restless extremity movements, verbal responses)
Severity of pain at suprapubic area | at 0, 1, 2, and 6 hours after extubation
  Pain at suprapubic area will be evaluated using VAS after extubation
Sedation level | at 0, 1, 2, and 6 hours after extubation
  The Ramsay Sedation Scale was measured
Incidence of treatment-emergent adverse events | at 0, 1, 2, and 6 hours after extubation
  The incidence of nausea, vomiting, hypotension, hypertension, bradycardia,respiratory depression after extubation, and excessive sedation were also recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Yang, PhD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No